CLINICAL TRIAL: NCT01954303
Title: Elevated High-sensitivity Cardiac Troponin T Levels in Patients With Stable Coronary Artery Disease
Brief Title: HsTnT in Stable Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Moritz Biener, Resident, University Hospital Heidelberg
Other Study IDs: UHHD-BM-001
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Troponin status: Patients are divided into "troponin positive" (if hsTnT on first presentation is <14 ng/L) and "troponin negative" (if hsTnT on first presentation is >=14 ng/l).
  Interventions: Other: Progress of CHD
- Progress of CHD

INTERVENTIONS:
Other: Progress of CHD
  Groups: Troponin status

SUMMARY:
Coronary artery disease (CAD) is one of the leading causes of morbidity and mortality worldwide. Life threatening manifestations such as acute myocardial infarction (AMI) and sudden cardiac death are the most important causes of death in many countries. Cardiac troponin is a biomarker with a high specificity for cardiac necrosis and is recommended for diagnosis of acute myocardial infarction by the Universal definition of myocardial infarction. Since a new generation of high-sensitivity cardiac troponin assays has become commercially available a few years ago, myocardial infarction can be detected earlier and even small AMIs, that were classified as unstable angina pectoris (UAP) with the less sensitive assays, are detectable now. On the other side, more patients with acute or chronic myocardial damage not due to AMI are identified now. Thereby, the reason for elevated troponin levels should be sought actively, because high troponin levels were associated with adverse outcome - independent of the underlying pathomechanism. The reasons for troponin elevations in patients with stable CAD are not clear yet. Associations with extensive atherosclerosis, carotid lesions and complex coronary plaques in coronary CT scans were reported. Therefore, patients with elevated troponin levels represent a risk population and might profit from intensified secondary prevention. In this context, ticagrelor might be part of a prevention strategy as currently tested in the PEGASUS trial.

We plan to conduct a single-centre pilot study in a cohort with clinically stable patients of our outpatient clinic, because data regarding prevalence, causes and prognosis of elevated troponin values in unselected cohorts is sparse. Therefore, all patients (n=910) that presented to our outpatient clinic 12 months after introduction of the high-sensitivity troponin T assay (june 2009) and were free of complaints or presented with UAP are being enrolled. All patients are characterized by demographic, laboratory and clinical characteristics (including medication) and all available imaging data (exercise-ecg, echocardiography, stress-echocardiography, computed tomography, cardiac MRI and coronary angiography) in order to compare baseline characteristics of troponin positive and troponin negative patients. In addition, the Framingham- and PROCAM-Score representing established calculators of long-term risk prediction are calculated.

Prognostic endpoints are defined as severe cardiovascular events and progress of the initially diagnosed disease. Those endpoints are associated with the initial hs-cTnT value and serial changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients of outpatient clinic presenting 12 months after introduction of the hs-TnT test in june 2009

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to conduct a single-centre pilot study in a cohort with clinically stable patients (n=910) of our outpatient clinic who presented 12 months after introduction of the high-sensitivity troponin T assay (june 2009) for routine workup. No patients will be excluded.
  All patients with stable CAD with or without cardiovascular comorbidities will be selected and classified as "troponin positive" or "troponin negative" according to initially documented hs-cTnT value.
Sampling Method: Non-Probability Sample
Enrollment: 965 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death | 3 years

SECONDARY OUTCOMES:
Recurrent Myocardial Infarction | 3 years

OTHER OUTCOMES:
Recurrent coronary intervention | 3 years

REFERENCES:
- [Derived] Biener M, Giannitsis E, Hogrefe K, Mueller-Hennessen M, Frohlich H, Katus HA, Frey N, Frankenstein L, Tager T. Prognostic value of changes in high-sensitivity cardiac troponin T beyond biological variation in stable outpatients with cardiovascular disease: a validation study. Clin Res Cardiol. 2022 Mar;111(3):333-342. doi: 10.1007/s00392-021-01952-6. Epub 2021 Oct 25. PMID 34694435
- [Derived] Tager T, Giannitsis E, Greve K, Frohlich H, Muller-Hennessen M, Vafaie M, Katus HA, Frankenstein L, Biener M. Long-term biological variation of high-sensitivity cardiac troponin T using minimal important differences and reference change values in stable outpatients with cardiovascular disease. Clin Biochem. 2019 May;67:7-11. doi: 10.1016/j.clinbiochem.2019.03.003. Epub 2019 Mar 11. PMID 30872042
- [Derived] Biener M, Giannitsis E, Kuhner M, Zelniker T, Mueller-Hennessen M, Vafaie M, Stoyanov KM, Neumann FJ, Katus HA, Hochholzer W, Valina CM. Risk prediction in stable cardiovascular disease using a high-sensitivity cardiac troponin T single biomarker strategy compared to the ESC-SCORE. Open Heart. 2018 Apr 25;5(1):e000710. doi: 10.1136/openhrt-2017-000710. eCollection 2018. PMID 29713483